CLINICAL TRIAL: NCT03019926
Title: Lupus and Observance
Acronym: LUPOBS
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 16/B/09
Record Dates: First submitted 2017-01-10; First posted 2017-01-13 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2018-06

CONDITIONS: Systemic Lupus, Skin Lupus
Keywords: systemic lupus erythematosus; observance; hydroxychloroquine dosage; risk factors of non-observance; SLICC score; SLEDAI score
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Hydroxychloroquine dosage — Blood sample from a 6 ml tube, performed in the common practice.

SUMMARY:
A poor therapeutic observance is described between 3 and 76% cases in systemic lupus. It is associated with an increased risk of relapses, hospitalizations, morbidity and poor renal prognosis.

New treatment protocols exist and are indicated in second intention in case of good compliance. An assessment of therapeutic adherence is therefore essential.

Patients with systemic lupus diagnosed for at least 6 months, or skin lupus, who have been prescribed with Plaquenil (hydroxychloroquine), will be included in the study.

The study primary objective is to determine risk factors for non-observance

The secondary objectives are to:

* Measure the observance rate of patients with systemic lupus in Martinique.
* Describe the parameters that influence observance: evaluation of the disease and associated comorbidities, psychosocial assessment, assessment of the doctor-patient relationship, evaluation of the disease representations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Systemic lupus defined according to the diagnostic criteria of the American College of Rheumatology " 1997, diagnosed for at least 6 months; Or Skin Lupus
3. Consultation or hospitalization at the University Hospital of Martinique, in either services of Internal Medicine, Rheumatology or Dermatology.
4. Prescription of hydroxychloroquine (Plaquenil®) for at least 6 months
5. Affiliate or beneficiary of a social security scheme.
6. Patient not opposed to participate in the study

Exclusion Criteria:

1. Age <18 years or patient under guardianship
2. Patient not speaking and / or not understanding French
3. No prescription and/or contraindication to hydroxychloroquine
4. Systemic lupus outbreak with neurological impairment defined by SLEDAI score by a psychosis (disruption of normal activity in relation to a severe alteration of the perception of reality. Includes: hallucinations, incoherence, impoverishment of the content of thought, illogical reasoning, bizarre behavior, disorganized or catatonic) or brain damage (with impairment of mental functions with impaired orientation, memory or other brutal appearance and fluctuating evolution).
5. History of psychiatric disorders: personality disorders, psychoses, severe depression
6. Hospitalization with a life-threatening clinical condition that does not allow to answer questions
7. Non affiliated patient or beneficiary of a social security scheme.
8. Patient refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will is proposed to anyone aged 18 years or older with a diagnosis of systemic lupus or skin lupus for at least 6 months, ans who has been prescribed with hydroxychloroquine (Plaquenil) for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is based on a blood dosage of hydroxychloroquine (HCQ) | Reflects the Plaquenil intake during the 40 previous days
  The HCQ dosage is assayed on whole blood (6ml) by high-pressure liquid chromatography performance, reproducible and inexpensive method. Only one laboratory centralizes the sampling.
  A dosage below 200 ng/ml or 0.2 mg/l defines a non-observing patient within the 40 days above.

SECONDARY OUTCOMES:
Patients considered as observing and non-observing will be compared according to the activity of the disease | 40 days
  Activity of the disease : Systemic lupus considered as active for a SELENA-SLEDAI score ≥ 6
Patients considered as observing and non-observing will be compared according to number of prescribed medication | 40 days
Patients considered as observing and non-observing will be compared according to the presence of anxiety and/or depressive disorders | 40 days
  Presence of anxiety and/or depressive disorders, according to the Hospital Anxiety And Depression Scale (HAD), a score > to 10

CONTACTS AND LOCATIONS:
Overall Officials: Katlyne POLOMAT, MD, Principal Investigator — CHU of Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique, France

IPD SHARING:
Plan to Share IPD: No